CLINICAL TRIAL: NCT03795844
Title: COMPARISON OF LIVER RETRACTOR USED IN LAPAROSCOPIC SLEEVE GASTRECTOMY BY INTRAOPERATIVE LIVER DAMAGE
Brief Title: COMPARISON OF LIVER RETRACTOR FOR INTRATOPERATIVE LIVER DAMAGE
Acronym: RETRACTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ANIL ERGIN, Dr Anil ERGIN , General Surgery , Asistant doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ANIL ERGIN.......
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Liver Damage

STUDY DESIGN:
Intervention Model Description: In this study, 120 patients who are over 18 years old with laparoscopic sleeve gastrectomy will be included. 4 groups will be formed and each group will be planned to include 30 patients. In group 1, a 5 mm incision was made under xiphoid during the operation, and Nathanson retractor was placed and liver left lobe retraction would be achieved. In the second group, a snake retractor with a 5 mm incision under the xiphoid will be used. In the 3rd group, liver retraction will be provided by using a 5 mm trocar from the intersection of the right midclavicular line. In the control group, liver retraction through a 5 mm trocar entrained from the intersection of the right midclavicular line and a 4 cm superior umbilicus will be provided with the aid of laparoscopic grasper without any special tools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nathanson retractor (Active Comparator): Liver retraction in group 1, a 5 mm incision was made under xiphoid during the operation, and Nathanson retractor was placed and liver left lobe retraction would be achieved.
  Interventions: Procedure: liver retraction Nathanson retractor
- snake retractor (Active Comparator): Liver retraction in group 2 ; 5 mm incision under the xiphoid will be used. Snake retractor was placed and liver left lobe retraction would be achieved.
  Interventions: Procedure: liver retraction snake retractor
- fan retractor (Active Comparator): Liver retraction in group 3 ; through a 5 mm trocar entrained from the intersection of the right midclavicular line and a 4 cm superior umbilicus
  Interventions: Procedure: liver retraction fan retractor
- CONTROL GROUP (Active Comparator): Liver retraction in group 4 ; through a 5 mm trocar entrained from the intersection of the right midclavicular line and a 4 cm superior umbilicus will be provided with the aid of laparoscopic grasper without any special tools
  Interventions: Procedure: liver retraction laparoscopic grasper

INTERVENTIONS:
Procedure: liver retraction Nathanson retractor — liver retractor will be used for the retraction of left lobe of liver
  Other Names: nathanson retractor
  Arms: Nathanson retractor
Procedure: liver retraction snake retractor — liver retractor will be used for the retraction of left lobe of liver
  Arms: snake retractor
Procedure: liver retraction fan retractor — liver retractor will be used for the retraction of left lobe of liver
  Arms: fan retractor
Procedure: liver retraction laparoscopic grasper — laparoscopic grasper without any special tools
  Arms: CONTROL GROUP

SUMMARY:
The frequency of laparoscopic bariatric surgery is increasing day by day. In these surgeries, the liver masses are also found to be significantly larger due to the high Body Mass Index scores. It is known that the application of a diet called liver shrinkage protein diet which is applied preoperatively is a method that contributes to the comfort of the surgeon during surgery by reducing the size of the liver. The large size of the liver narrows the field of view of the surgeon in operation and decreases the comfort of surgery. One of the most important points that the surgeon must solve during surgery is the exclusion of the left lobe of the liver. The most commonly used types of liver retractors today; Nathanson retractor, Snowden-Window retractor, Snake retractor, Fan retractor, LIvac retractor and many other retractors. Some of these retractors require an additional incision under xiphoid, which may lead to an injury risk. The installation of these retractors also increases the operation time and requires additional time. Numerous studies have shown that retractors, which are used to rule out liver left lobe during surgery, cause liver damage. However, in order to reveal His angle in the esophageal-gastric composition, hepatic left lobe exclusion is mandatory. Therefore, it is necessary to determine and use the retractor type which causes the least damage between the liver retractors. In our study, it was aimed to reveal three types of liver retractors in our hospital in different cases and to reveal the type of trocar that causes the least amount of liver damage.

DETAILED DESCRIPTION:
During laparoscopic upper abdominal surgery, the operative view is usually blocked by the left lobe of the liver. An effective liver retraction is important for good vision and safety during operation. In this study, 120 patients who are over 18 years old with laparoscopic sleeve gastrectomy will be included. 4 groups will be formed and each group will be planned to include 30 patients. In group 1, a 5 mm incision was made under xiphoid during the operation, and Nathanson retractor was placed and liver left lobe retraction would be achieved. In the second group, a snake retractor with a 5 mm incision under the xiphoid will be used. In the 3rd group, liver retraction will be provided by using a 5 mm trocar from the intersection of the right midclavicular line. In the group, liver retraction through a 5 mm trocar entrained from the intersection of the right midclavicular line and a 4 cm superior umbilicus will be provided with the aid of laparoscopic grasper without any special tools. In these patients, aspartate aminotransferase, alanine aminotransferase and Bilirubin levels will be examined on the postoperative 1st, 2nd and 3rd days and the patients will be examined with postoperative first day abdominal abdomen magnetic resonance imaging and the liver injury will be evaluated by the radiologist. Patients will not know which liver excision method is used during surgery. The radiologist who will perform damage assessment on imaging will not know which type of liver dislocation is used. Therefore, the study will be planned as double blind. The liver excision method will be applied sequentially. Randomization will be done in this way.

ELIGIBILITY:
Inclusion Criteria:

* The patients older than 18 years planned for Laparoscopic Sleeve Gastrectomy

Exclusion Criteria:

* The patients with liver failure
* The patients with impaired preoperative liver function tests
* The patients who have been diagnosed with any liver disease
* The patients with bleeding disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Liver damage of liver retractors by measurement of AST(Aspartate Aminotransferase), ALT (alanine aminotransferase) , GGT (Gamma-Glutamyl Transferase) , Bilirubin (Total , direct , indirect ) levels. | 72 hours
  measurement of AST(Aspartate Aminotransferase), ALT (alanine aminotransferase) , GGT (Gamma-Glutamyl Transferase) , Bilirubin (Total , direct , indirect ) levels will be measured preoperatively and postoperative 0 , 1 , 2 , 3 days and record.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No